CLINICAL TRIAL: NCT04833153
Title: Continuing Education Intervention "Person First - Please" of Person-Centred Care Targeted to Nurses in Older People Long-term Care
Brief Title: Continuing Education Intervention Named "Person First - Please"
Acronym: PFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mari Pakkonen (Other)
Responsible Party: Sponsor-Investigator, Mari Pakkonen, PhD-candidate, University of Turku
Organization: University of Turku (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: mjpakk73645
Record Dates: First submitted 2021-03-13; First posted 2021-04-06 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Nurse-Patient Relations
Keywords: Person-centred care; Continuing education; Long-term care; Older people

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFP intervention (Experimental): PFP 10 week continuing education intervention
  Interventions: Behavioral: Person-First - Please (PFP)
- Control arm (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Person-First - Please (PFP) — PFP takes 10 weeks and consist of four modules: Information, Person, Autonomy and Dignity. Information module takes 1 hour contact on first week. The other modules will follow every third weeks, starting from week 2. So that on week 2, 5 and 8 researcher meet nurses in 4 hours education session. Between the modules, nurses can take contact online to the researcher.
  Arms: PFP intervention

SUMMARY:
The aim of this study is to evaluate the effectiveness of the Person-First - Please (PFP) intervention in supporting nurse's competence and collective competence of Person-Centred Care (PCC) in older people Long-Term Care (LTC). The goal is to promote PCC culture in older people LTC.

Research question 1:

What is the effectiveness of the PFP intervention on the PCC collective competency of nurses in older people LTC?

Hypothesis for research question 1 are:

1. Nurses in intervention group will have higher level of competence of PCC than control.

Research question 2:

How PCC climate has been maintained in older people LTC from the point of view of the nurses, next of kin and older people?

Hypothesis for research question 2 are:

1. PCC climate will be better in intervention group than control from point of view of the nurses, next of kin and older people.
2. The higher competence of nurses the higher level of PCC climate from point of view of the next of kin and older people.
3. The higher collective competence of the nurses the higher level of the PCC climate from point of view of the next of kin and older people.

DETAILED DESCRIPTION:
The study takes place in older people long-term care on two cities in western part of Finland. The long-term care units are similar as stuff structure, nurse/resident ration, working ideology and quality management.

The research design is quasi-experimental research with pre- and post- test measurements in the intervention and control groups. The intervention group will follow the protocol and the control group participants will follow the usually care. Data are being collected at baseline, immediately after 10 weeks intervention and at follow-up 6 weeks after intervention.

Continuing education named "Person First - Please" (PFP) based on Person-Centered Care (PCC) Practice Framework and Theory of Collective Competence and it consist of four modules: Information, Person, Autonomy and Dignity. Information module will take one hour in the first intervention week, and it will include information about the study; informed consent; short clarification about concept PCC and prerequisites for PCC. Tree other modules takes 4 hours contact with researcher in every three weeks.

Power analyses for the sample size showed that for 0.8 effect size, power of 0.8 and statistical significance of 0.05 with three main hypotheses, for intervention group n=64 and for control group n=128. ICC of 0.1 was used based on previous sample of the primary outcome measurement.

The sampling based on cluster sampling. Two cities will be constituting the clusters in western part of Finland. From these cities will be selected first all public long-term care units for the older people. To avoid contamination, one of the cities will be selected to participate in the intervention and the other in the control.

Participants in the study consist of nurses (Registered Nurses, Licensed Practice Nurses, Caregiver Assistants) who work in older people LTC and older people from the same units participate alone or with their next of kin.

Nurses background questions are age, education, working experience. Older people and next of kin background questions are age, length of the living in LTC, relationship, number of visits per week in LTC. The effectiveness of an intervention is measured by validated measurements that have been properly licensed.

The data will be analysed by latest version of the Software Platform for Statistical Analysis (SPSS). Descriptive statistic will be calculated for the numerical and categorical data. The normal distribution of the data and 95% confidence intervals will be calculated for the numerical and categorical data. Intervention and control group will be statistically compared, and differences will be measured at each time point. At the baseline will be ensure the similarity of intervention and control group for background variables. Cross-tabulations will be done for categorical and numerical variables. The sum variable of the measurements during the three different measurement time will be analysed using hierarchical linear mixed models will compare the changes over time between the groups.

Each participant will be informed before about the purpose of the study, issues related to research ethics, reporting of the findings and they will sign informed consent. Since the study involves research participants who are vulnerable due to cognitive impairment, researcher have clear protocol and special attention will be paid to ethical issues during the study.

ELIGIBILITY:
Inclusion Criteria:

* Nurses (RNs, Licensed Practice Nurses, Caregiver Assistants) who works in older people LTC. The inclusion criteria for nurses are that they work permanently or on a long-term deputy (at least 6 months) in units.
* The criteria for older people participating alone are that older people have enough cognitive capacity assessed by managers of the units. The criteria for next of kin participating is they will visit at least weekly in LTC.

Exclusion Criteria:

* short- time deputy nurses
* older people in terminal care

Max Age: 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in nurses PCC competency | baseline - after the intervention - 6 week follow up
  The competence data will be collected by the Patient-centred Care Competency (PCC) scale as primary outcome. The PCC scale consists of 17 items with 5-point Likert scale (1 = minimal, 2 = below average, 3 = average, 4 = good, 5 = excellent), divided subscales: respecting patients' perspectives, promoting patient involvement in care processes, providing for patient comfort, and advocating for patients.

SECONDARY OUTCOMES:
Changes in PCC climate in lens of nurses, older people and next of kin | baseline - after the intervention - 6 week follow up
  The PCC climate data will be collected by Person-centred questionnaire (PCQ-S) staff version and (PCQ-P) patient version (6- point Likert scale: 0 = No, I disagree completely; 1 = No, I disagree; 2 = No, I partly disagree, 3 = Yes, I partly agree; 4 = Yes, I agree; 5 = Yes, I agree completely). Scales are divided subscales: hospitality, safety and everydayness. Data will be collect from nurses, older people and their next of kin.
Evaluation of the continuing education named PFP in lens of the nurses | during the intervention
  A feasibility tool has been developed for this intervention. Data will be collected from the nurses in end of the every PFP-modules, excluded information module.
  Tool consist of the subscales: content of the PFP; evaluation about the pedagogical methods; utilization of the PFP; evaluation of the PFP dosage; evaluation of the trainer. There is 5-point Likert scale: 1 = disagree; 2 = partly disagree; 3 = no disagree/no agree; 4 = agree; 5 = agree completely.

CONTACTS AND LOCATIONS:
Overall Officials: Suhonen, Professor, Study Director — University of Turku
Locations (1):
- Social services and health care, Rauma, Satakunta, Finland

IPD SHARING:
Plan to Share IPD: No
small sample size and vulnerable participants

REFERENCES:
- [Derived] Pakkonen M, Stolt M, Edvardsson D, Pasanen M, Suhonen R. Person-centred care competence and person-centred care climate described by nurses in older people's long-term care-A cross-sectional survey. Int J Older People Nurs. 2023 May;18(3):e12532. doi: 10.1111/opn.12532. Epub 2023 Mar 14. PMID 36918384